CLINICAL TRIAL: NCT06249568
Title: Evaluation of Fluid Responsiveness With Recruitment Maneuver After Sternotomy in Coronary Artery Bypass Surgery
Acronym: fluidresponse
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Meltem Sakman Yılmaz, assistant doctor, Ankara City Hospital Bilkent
Other Study IDs: E2-23-3460
Record Dates: First submitted 2024-01-13; First posted 2024-02-08 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Fluid Therapy; Coronary Artery Bypass Surgery Patients; Lung Recruitment Maneuver
Keywords: fluid therapy; Coronary Artery Bypass Surgery Patients; Lung Recruitment Maneuver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who will have coroner arter bypass surgeon: Patients undergoing coronary artery bypass surgery will be eliminated if there are exclusion criteria. Patients who do not have exclusion criteria will be included in the study if they agree to volunteer.

SUMMARY:
Assuming that the basic reliability of dynamic indices will increase with the application of functional hemodynamic tests after sternotomy and protective lung ventilation in patients undergoing elective coronary artery bypass surgery, it is useful to predict fluid responsiveness after sternotomy in coronary artery bypass surgery patients ventilated with 6 ml/kg PBW (ideal body weight). We aimed to reveal the sensitivity and specificity of PPV and SVV changes by applying a lung opening maneuver.

DETAILED DESCRIPTION:
In order to evaluate the fluid deficit in patients undergoing coronary artery bypass surgery, researchers will measure stroke volume index, cardiac index and mean arterial pressure while the patients are in the lima position.

Then researchers will perform a lung opening maneuver (30mmHg for 30 seconds) and measure again.

researchers will measure again after the values return to normal. researchers will give patients balanced fluid at 3ml/kg and record their values.

Can researchers predict fluid response with lung opening maneuver?

ELIGIBILITY:
* Inclusion Criteria:
* 1-ASA2-3 patients between the ages of 18-80 who will undergo elective coronary bypass surgery under general anesthesia
* Exclusion Criteria:
* 1. Be younger than 18 years old, be over 80 years old
* 2. Patients with an ASA score greater than 3
* 3. EF<40%
* 4. Those with contraindications to anesthetic drugs
* 5. Patients with BMI>30
* 6. Patients who did not want to participate in the study
* 7. Right ventricular dysfunction
* 8. COPD(Chronic obstructive pulmonary disease)
* 9. Bullous lung disease
* 10. Moderate to severe PHT
* 11. Severe kidney or liver disease
* 12. Patients with hemodynamic instability in the perioperative period
* 13. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA2-3 patients between the ages of 18-80 who will undergo elective coronary bypass surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-02 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Determination of fluid responsiveness in patients undergoing coronary arter bypass surgery. | from start to 4 months
  : Demonstration of fluid responsiveness in patients who will undergo coronary artery bypass surgery will prevent unnecessary fluid administration in case of hemodynamic disturbance, and medical treatments and interventions can be performed in a timely and targeted manner. Researchers will perform a recruitment maneuver on the patients and record mean arterial pressure and stroke volume index.
  Researchers will perform a recruitment maneuver on the patients and record mean arterial pressure and stroke volume index.
  Afterwards, researchers will give 3ml/cc balanced fluid to the patient and record the change in mean arterial pressure and stroke volume index.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
fluid responsiveness